CLINICAL TRIAL: NCT04580888
Title: Impact of Early Haemodynamic Assessment by Echocardiography on Organ Dysfunction of Patients Admitted in the Emergency Department for Sepsis or Septic Shock
Brief Title: Emergency Echocardiography in Sepsis
Acronym: GENESIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87RI19_0038 (GENESIS)
Record Dates: First submitted 2020-09-28; First posted 2020-10-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Echocardiography; Organ Dysfunction Syndrome Sepsis; Emergencies
Keywords: Sepsis; Echocardiography; Haemodynamic; Emergency Medicine
MeSH Terms: conditions — Sepsis; Toxemia; Emergencies | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Assessment using an early transthoracic echocardiography (after 500 mL of fluids) to identify the hemodynamic profile responsible for the acute circulatory failure associated with sepsis / septic shock and to guide ongoing treatment (therapeutic algorithm) and monitor its efficacy and tolerance.
  Interventions: Procedure: early transthoracic echocardiography
- Control arm (Other): Conventional management according to current standards of care based on SSC recommendations, including a standardized fluid resuscitation of 30 mL/kg.
  Interventions: Procedure: standards of care

INTERVENTIONS:
Procedure: early transthoracic echocardiography — In the intervention arm, echocardiography will be performed immediately and potentially repeated to confirm the need for additional fluid resuscitation up to 30 mL/kg in the presence of persisting hypovolemia, or not (e.g., severe ventricular dysfunction). A therapeutic algorithm will allow standardized impact on ongoing management according to the hemodynamic profile identified by early echocardiography. After the completion of initial fluid resuscitation up to 30 mL/kg if required, a new echocardiographic assessment will be systematically performed by the same operator to stop or not fluid resuscitation, and to potentially initiate another treatment according to both the hemodynamic profile and clinical context.
  Arms: Intervention arm
Procedure: standards of care — In the control arm, patients will be treated according to standards of care based on current SSC recommendations, including a fluid resuscitation of 30 mL/kg.
  Arms: Control arm

SUMMARY:
Acute circulatory failure that combines hypovolemia, vasoplegia and cardiac dysfunction plays a major role in the development of sepsis-related organ dysfunction. Pathophysiological mechanisms are multiple and complex. The objective of the GENESIS study is to determine the impact of early haemodynamic assessment using echocardiography in association with a therapeutic algorithm (intervention arm), when compared with standard of care based on the current Surviving Sepsis Campaign (SSC) recommendations (control arm), on the development of organ dysfunctions in patients admitted to the Emergency Department for sepsis or septic shock.

DETAILED DESCRIPTION:
Sepsis is currently defined as life-threatening organ dysfunction secondary to a dysregulated host response to infection (Sepsis-3). Septic shock is a subgroup of patients who also have sustained arterial hypotension requiring vasopressors and tissue dysoxia. The mortality varies from 10 to 40% depending on the severity. The latest "bundles" of the SSC request to perform within the first hour of sepsis identification a fluid loading of 30 mL/kg of crystalloids in the presence of hypotension, and to initiate a vasopressor support in case of persistent hypotension to maintain a mean arterial pressure ≥ 65 mmHg. However, early fluid resuscitation is not necessarily associated with an improvement of sepsis prognosis and may even be deleterious when leading to excessive positive fluid balance. Accordingly, the SSC recommends investigating a personalized approach to define for each patient the appropriate volume of fluids to be administered according to the initial mechanism of sepsis-induced cardiovascular failure. Echocardiography is currently recommended as a first-line modality to identify the origin of acute circulatory failure, sepsis remaining the leading cause. It has been shown to alter ongoing treatment based on the sole SSC recommendations in the intensive care unit. In contrast, the impact of hemodynamic assessment using echocardiography at the early stage of sepsis in patients admitted to the Emergency Department (ED) is unknown.

In this randomized trial, patients will be either assessed hemodynamically using transthoracic echocardiography to guide early therapeutic management (intervention arm) or managed according to standards of care based on current SSC recommendations (control arm). Early echocardiography will be performed after 500 mL of fluid loading initiated upon identification of septic patients based on the qSOFA score (hemodynamic criterion required: systolic blood pressure ≤ 100 mmHg). This will allow identifying the hemodynamic profile at the origin of sepsis-induced circulatory failure and to monitor both the efficacy and tolerance of fluid resuscitation, or of any other therapeutic intervention (e.g., inotropic support) according to a predefined therapeutic algorithm. Patients allocated to the control arm will be managed conventionally according to current SSC recommendations, including a standardized fluid loading of 30 mL/kg.

Organ dysfunctions will be assessed in the two study arms by the SOFA score 24 hours after randomization and patient will be followed up until hospital discharge to determine outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ED
* Age ≥ 18 years and affiliation to Social Security
* With sepsis (Sepsis-3 definition):

Clinically suspected or documented acute infection

AND a quick score Sequential Organ Failure Assessment (qSOFA) ≥ 2 points with:

* Systolic blood pressure ≤ 100 mmHg (1 point) requiring fluid loading
* AND encephalopathy (1 point) OR respiratory rate ≥ 22 cpm (1 point) AND a systolic blood pressure ≤ 100 mmHg after 500 mL of crystalloid vascular filling - Informed consent

Exclusion Criteria:

* Decision to limit care or moribund status
* Pregnancy or breast feeding
* Subject under juridical protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Change in Sequential Organ Failure Assessment (SOFA) score | change from Hour 0 at Day 1
  Crude variation of the SOFA score between inclusion and 24h following randomization.

SECONDARY OUTCOMES:
Interruption of fluid resuscitation | Hour 3
  Number and proportion of patients in whom echocardiography performed in the ED (intervention arm) modified ongoing therapy based on SSC recommendations (standard of care) according to the hemodynamic profile. Interruption of fluid resuscitation before having administrated 30 mL/kg
Maintains of fluid resuscitation | Hour 3
  Number and proportion of patients in whom echocardiography performed in the ED (intervention arm) modified ongoing therapy based on SSC recommendations (standard of care) according to the hemodynamic profile. Fluid resuscitation maintained beyond 30 mL/kg
Initiation of inotropes | Hour 3
  Number and proportion of patients in whom echocardiography performed in the ED (intervention arm) modified ongoing therapy based on SSC recommendations (standard of care) according to the hemodynamic profile. Initiation of inotropes
Initiation of vasopressor support | Hour 3
  Number and proportion of patients in whom echocardiography performed in the ED (intervention arm) modified ongoing therapy based on SSC recommendations (standard of care) according to the hemodynamic profile. Initiation of vasopressor support
Therapeutic modification | Hour 3
  Number and proportion of patients in whom echocardiography performed in the ED (intervention arm) modified ongoing therapy based on SSC recommendations (standard of care) according to the hemodynamic profile. Therapeutic modification directly related to the echocardiographic examination
Persisting hypovolemia | Hour 0
  Number and proportion of patients presenting at the time of early hemodynamic assessment using echocardiography (intervention arm)
Left ventricular failure | Hour 0
  Number and proportion of patients presenting at the time of early hemodynamic assessment using echocardiography (intervention arm)
Vasoplegia with left ventricular hyperkinesia | Hour 0
  Number and proportion of patients presenting at the time of early hemodynamic assessment using echocardiography (intervention arm)
Right ventricular failure | Hour 0
  Number and proportion of patients presenting at the time of early hemodynamic assessment using echocardiography (intervention arm)
Stabilized hemodynamic status | Hour 0
  Number and proportion of patients presenting at the time of early hemodynamic assessment using echocardiography (intervention arm). Stabilized hemodynamic status (none of above-mentioned abnormalities) due to adequate management of acute circulatory failure (avoid any deleterious therapeutic change).
Hydrostatic pulmonary edema | through study completion, an average of 1 month
  Number of Hydrostatic pulmonary edema (cardiogenic or volume overload) since potentially related to excessive fluid loading
Supraventricular arrhythmias | through study completion, an average of 1 month
  Number of Supraventricular arrhythmias since potentially related to the initiation of positive inotropes
ventricular arrhythmias | through study completion, an average of 1 month
  Number of ventricular arrhythmias since potentially related to the initiation of positive inotropes
acute coronary syndrome, | through study completion, an average of 1 month
  Number of acute coronary syndrome since potentially related to the initiation of positive inotropes
ischemic stroke | through study completion, an average of 1 month
  Number of ischemic stroke since potentially related to the initiation of positive inotropes
hemorrhagic stroke | through study completion, an average of 1 month
  Number of hemorrhagic stroke since potentially related to the initiation of positive inotropes
Lactate clearance | Hour 0 to Hour 6
  Lactate clearance (lactate 6h after randomization compared to lactate at baseline)
septic shock | Hour 24
  Number and proportion of patients who developed septic shock 24 h after inclusion
Patient course | through study completion, an average of 1 month
  Patient course after emergency department discharge: hospitalization in regular ward (medicine / surgery), stepdown unit or intensive care unit.
Mortality | Day 7 and through study completion, an average of 1 month
  Mortality (all-cause and sepsis-related) at Day 7 and at hospital discharge

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CH d'Albi, Albi
  - CH d'Eaubonne - Montmorency, Eaubonne
  - Grenoble university hospital, La Tronche
  - Limgoes university hospital, Limoges
  - Hospices civils de Lyon, Lyon
  - Nantes university hospital, Nantes
  - Nice university hospital, Nice
  - Poitiers university hospital, Poitiers
  - La réunion university hospital, Saint-Pierre
  - Toulouse university hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided
The dataset generated and/or analysed during the current study will be made available from the principal investigator on reasonable request. The conditions for the transfer of all or part of the database will be decided by the study sponsor and will be the subject of a written contract.

REFERENCES:
- [Derived] Lafon T, Le Gouge A, Brit S, Giraudeau B, Vignon P. Impact of early haemodynamic assessment by echocardiography on organ dysfunction and outcome of patients admitted to the emergency department with sepsis or septic shock: protocol of a multicentre randomised controlled trial (GENESIS). BMJ Open. 2025 May 6;15(5):e098304. doi: 10.1136/bmjopen-2024-098304. PMID 40335132